CLINICAL TRIAL: NCT05044598
Title: RAFT - First in Human Phase I/II Clinical Trial of RAFT for Aniridia Related Keratopathy
Brief Title: RAFT - Clinical Trial of RAFT for Aniridia Related Keratopathy
Acronym: RAFT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Medical Research Council (Other Government); Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTU/2017/307
Record Dates: First submitted 2021-05-19; First posted 2021-09-16 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Aniridia
MeSH Terms: conditions — Aniridia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RAFT-OS (Other): Single-arm trial is to investigate if RAFT-OS ((Real Architecture for 3D Tissues Ocular Surface) is a safe and effective alternative treatment for patients with aniridia related keratopathy (ARK) in 21 patients.
  The RAFT-OS will be transplanted into the participants worst affected eye. Following surgery, each participant will be assessed at days 1, 7, 14, 21, and 1-month for major or intermediate safety events. Participants will continue to be followed up to 12 months after transplantation and will be required to stay on the immune suppression therapy for the duration of the trial.
  Interventions: Other: RAFT-OS

INTERVENTIONS:
Other: RAFT-OS — RAFT-OS (Real Architecture for 3D Tissues Ocular Surface) is an artificial tissue, populated with limbal epithelial cells and stromal cells.

SUMMARY:
The RAFT trial is a first in human trial of a novel cellular therapy called RAFT-OS (Real Architecture for 3D Tissues Ocular Surface) developed and manufactured by Cells for Sight Stem Cell Therapy Research Unit at UCL institute of Ophthalmology.

The aim of this seamless phase I/II single-dose, single-arm trial is to investigate if RAFT-OS is a safe and effective alternative treatment for patients with aniridia related keratopathy (ARK) in 21 patients.

ARK is a complication of aniridia, which is a genetic eye condition present from birth.

RAFT-OS is an artificial tissue, populated with limbal epithelial cells and stromal cells. The source of the adult limbal and stromal cells is from donated human corneas from the NHS blood and Transplant, Tissue and Eye services in Liverpool.

Following a Screening visit, participants will commence 10-weeks of immune suppression therapy to prepare for the transplantation of RAFT-OS.

The RAFT-OS will be transplanted into the participants worst affected eye. Following surgery, each participant will be assessed at days 1, 7, 14, 21, and 1-month for major or intermediate safety events. Participants will continue to be followed up to 12 months after transplantation and will be required to stay on the immune suppression therapy for the duration of the trial.

The trial is conducted at Moorfields Eye Hospital NHS Foundation Trust (MEH), London in the United Kingdom (UK). MEH is a leading provider of eye health services in the UK and is a world-class centre of excellence for ophthalmic research and education.

All trial medical assessments and procedures will be performed in an appropriate clinical setting by suitability qualified staff.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of congenital aniridia
2. Confirmed diagnosis of advanced aniridia related keratopathy with corneal surface conjunctivalisation, vascularisation and increasing opacity with worsening vision loss, glare & ocular surface pain
3. Patients aged 18 years and over
4. Participants must use acceptable contraception from enrolment up to 6 weeks for female participants and 90 days for male participants, after stopping immunosuppression therapy
5. Negative viral screen for, HIV, syphilis, hepatitis B & C and Human T-cell Leukaemia Virus (HTLV)
6. Negative urine pregnancy test.

Exclusion Criteria:

1. Poor tear production, as assessed by a Schirmer's test type 1
2. Lid malposition (entropion, ectropion, fornix shortening, symblepharon)
3. Current corneal infection
4. Uncontrolled glaucoma (defined as uncontrolled eye pressure, changes to medication, recent surgery in the last 3 months or being considered for surgical treatment)
5. Must not be NPL (no light perception) in one or both eyes
6. Patients who refuse to consent to the site informing their GP of their participation
7. Patients who lack capacity to give full informed consent to participate
8. Pregnant or lactating women
9. Patients with known contraindications to any of the following non-investigational medicinal products; mycophenolate, prednisolone, omeprazole, doxycycline, dexamethasone & moxifloxacin or excipients according to the relevant SmPCs
10. Patients who are participating in any concurrent trial involving an investigational medical product, device or surgical intervention within the last 12 months
11. Known albumin or egg allergy
12. Known penicillin allergy
13. Known hydrocortisone allergy
14. Inability to lie flat for surgical procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2025-04-17 (Actual); Study Completion 2025-04-17 (Actual)

PRIMARY OUTCOMES:
Primary safety outcome defined as the number of adverse events related to the intervention | 12 months
  defined as either major adverse event (non-ocular SUSAR; corneal melting; death) or any intermediate adverse event (persisting epithelial defect; persisting ocular inflammation; loss of corneal clarity; ocular SAEs related to the RAFT-OS and not surgery alone, conjunctival or lid swelling considered related to the ATIMP (RAFT-OS) and not surgery alone).
primary efficacy outcome defined as Improvement in the corneal surface at 3months post intervention. | 3 months
  Efficacy will be based on corneal surface normalisation (i.e., persistence of normal corneal epithelium and absence of vascularisation, epithelial defect and conjunctivalisation) at 3 months post-RAFT-OS transplantation using a validated ocular surface scoring system

SECONDARY OUTCOMES:
Change in visual acuity | 3 & 12 months post RAFT transplantation
  1. Visual improvement assessed by distance EDTRS visual acuity (refractive best corrected) at 3 & 12 months post RAFT-OS transplantation.
changes in quality of life scores | at 3 & 12 months post RAFT transplantation
  as assessed by NEI-VFQ-25 patient questionnaire
Changes in quality of Life scores | 3 &12 months post RAFT transplantation.
  RAND 36-Item Health Survey.

CONTACTS AND LOCATIONS:
Overall Officials: Sajjad Ahmad, Principal Investigator — Moorfields Eye Hospital, London; Julie Daniels, Study Chair — University College, London
Locations (1):
- Moorfields Eye Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No